CLINICAL TRIAL: NCT02793505
Title: Pregnancy Outcome Following Maternal Exposure to Metformin: a Collaborative ENTIS Study
Brief Title: Safety of Metformin in Pregnancy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Alice Panchaud, Senior research associate, Centre Hospitalier Universitaire Vaudois
Other Study IDs: STIS-05
Record Dates: First submitted 2016-05-25; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Pregnancy; Pregestational Diabetes; Polycystic Ovary Syndrom
Keywords: metformin; pregnancy outcomes; birth defects; spontaneous abortion; pharmacoepidemiology
MeSH Terms: conditions — Congenital Abnormalities; Abortion, Spontaneous | interventions — Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Pregnant patient exposed to metformin: Pregnant women seeking counseling by themselves or through their healthcare provider for exposure to metformin (Anatomical Therapeutic Chemical A10BA02) any time during pregnancy (i. e. any time from conception to week 42 after last menstrual period (LMP)).
  Interventions: Drug: metformin
- Reference group: Pregnant women seeking counseling by themselves or through their healthcare provider for exposure to any drug not known as a major teratogen or fetotoxicant and different than metformin, insulin or any other hypoglycaemic agent.
  Interventions: Drug: any drug not known as a major teratogen or major fetotoxicant

INTERVENTIONS:
Drug: metformin — This is not an intervention but an observed exposure.
  Groups: Pregnant patient exposed to metformin
Drug: any drug not known as a major teratogen or major fetotoxicant — This is not an intervention but an observed exposure.
  Groups: Reference group

SUMMARY:
This study aims to better characterize the risk linked to metformin use during pregnancy, using a prospective multicentric cohort design enabling a large sample size, in evaluating the rate of birth defects after first trimester exposure, as well as several other pregnancy related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Exposed group: exposed to metformin (Anatomical Therapeutic Chemical A10BA02) any time during pregnancy (i. e. any time from conception to week 42 after last menstrual period (LMP)).
* Reference group: at no time during pregnancy were exposed to metformin, insulin or any other hypoglycaemic agent.

Exclusion Criteria:

* exposed to any of the following known major teratogen or major fetotoxicant: acitretin, isotretinoin, mycophenolate, thalidomide, valproic acid, angiotensin-II receptor blockers (only when used in 2nd or 3rd trimester), ACE inhibitors (only when used in 2nd or 3rd trimester), or (b) following treatment indications coded: malignancies (MedDRA code: malignant or unspecified tumors (SMQ 20000091), ICD-10: C00-D09)) or malignancy related conditions (MedDRA: SMQ 20000092), ICD-10: C00-D09).
* lost to follow-up

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient from the European Network of Teratology Information Services (ENTIS) Cohort. This cohort is composed with patients, seeking counseling on the safety and risks regarding medication exposures in the reproductive age by themselves or through their healthcare provider. Each center gathers structured information on the exposure (medication, time of exposure, dose), maternal demographics, as well as medical and obstetric histories is collected prospectively. After the estimated date of birth, follow-up information on pregnancy outcome, gestational age at delivery, birth weight, congenital anomalies and neonatal complications is gathered through structured telephone interviews and/or mailed questionnaires sent to the mothers or their healthcare providers.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Major birth defects | within two weeks after birth or at histopathological exam in case of late spontaneous abortion or stillbirth occuring in pregnancy
Spontaneous abortion | until 20 weeks of pregnancy

SECONDARY OUTCOMES:
Minor birth defects | within two weeks after birth
Preterm birth | after 24 weeks of pregnancy
Pregnancy complications | after 12 weeks of pregnancy until delivery